CLINICAL TRIAL: NCT02618083
Title: Prognostic Value of Hemodynamic Disturbances of the Central Retinal Artery in Color Doppler Ultrasound in Rhegmatogenous Retinal Detachment
Brief Title: Prognostic Value of Hemodynamic Disturbances in Rhegmatogenous Retinal Detachment (CRADO-RED)
Acronym: CRADO-RED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALR_2015_24
Record Dates: First submitted 2015-11-26; First posted 2015-12-01 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- retinal detachment (Experimental): color Doppler ultrasound of the eye
  Interventions: Device: color Doppler ultrasound

INTERVENTIONS:
Device: color Doppler ultrasound — pre-operative blood flow velocity measurement with a color Doppler ultrasound device

SUMMARY:
Retinal detachments correspond to a separation of the neuroepithelium from the pigment epithelium. They can be exudative (sometimes in conjunction with a tumor), tractional, traumatic (postoperative) or rhegmatogenous (in relation to a tear).

Ultrasound, requested when the fundus is difficult to achieve and shows a hyperechoic mobile membrane. It can also measure the hemodynamic parameters of retinal arteries.

A preliminary study showed a correlation between systolic velocity in the central retinal artery and postoperative visual acuity.

The aim of this study is to confirm those preliminary data.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* rhegmatogenous retinal detachment, relapsing or not, including pseudophakic retinal detachment or aphakic retinal detachment, if the retinal detachment occurs more than three months after phacoemulsification

Exclusion Criteria:

* traumatic retinal detachment
* bilateral retinal detachment
* less than 3 months after phakoemulsification
* predictable follow-up of less than 6 months
* patient under of legal protection
* patient's opposition to participate
* absence of affiliation to the social security
* eye's axial length> 25.5 mm
* preoperative visual acuity greater than 70/100
* no surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity measured with the Early Treatment Diabetic Retinopathy Study (ETDRS) scale before surgery and at the sixth week of follow-up | Six weeks

SECONDARY OUTCOMES:
Visual acuity measured with the Early Treatment Diabetic Retinopathy Study (ETDRS) scale before surgery and at the sixth :month of follow-up | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France